CLINICAL TRIAL: NCT03332784
Title: A Phase 1 Study of TAK-925 to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Dose of TAK-925 in Healthy Adult and Elderly Volunteers and Patients With Narcolepsy
Brief Title: Phase 1 TAK-925 Study in Healthy Adult and Elderly Volunteers and Participants With Narcolepsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: TAK-925-1001; U1111-1201-6634 (Other: WHO); JapicCTI-173756 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Results first posted 2020-11-18 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Healthy Participants and Patients With Narcolepsy
MeSH Terms: interventions — TAK-925

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Part 1: TAK-925 (Cohort 1; Dose Level 1) (Experimental): TAK-925, Intravenous single administration. Healthy adults will be enrolled in double blind manner.
  Interventions: Drug: TAK-925
- Part 1: TAK-925 (Cohort 2; Dose Level 2) (Experimental): TAK-925, Intravenous single administration. Dose level will be determined by targeted plasma level of TAK-925 (Dose level 2). Dose selected based on safety, tolerability and PK data from previous Cohorts. Healthy adults will be enrolled in double blind manner.
  Interventions: Drug: TAK-925
- Part 1: TAK-925 (Cohort 1; Dose Level 3) (Experimental): TAK-925, Intravenous single administration. Dose level will be determined by targeted plasma level of TAK-925 (Dose level 3). Dose selected based on safety, tolerability and PK data from previous Cohorts. Healthy adults will be enrolled in double blind manner.
  Interventions: Drug: TAK-925
- Part 1: TAK-925 (Cohort 2; Dose Level 4) (Experimental): TAK-925, Intravenous single administration. Dose level will be determined by targeted plasma level of TAK-925 (Dose level 4). Dose selected based on safety, tolerability and PK data from previous Cohorts. Healthy adults will be enrolled in double blind manner.
  Interventions: Drug: TAK-925
- Part 1: TAK-925 (Cohort 1; Dose Level 5) (Experimental): TAK-925, Intravenous single administration. Dose level will be determined by targeted plasma level of TAK-925 (Dose level 5). Dose selected based on safety, tolerability and PK data from previous Cohorts. Healthy adults will be enrolled in double blind manner.
  Interventions: Drug: TAK-925
- Part 1: TAK-925 (Cohort 2; Dose Level 6) (Experimental): TAK-925, Intravenous single administration. Dose level will be determined by targeted plasma level of TAK-925 (Dose level 6). Dose selected based on safety, tolerability and PK data from previous Cohorts. Healthy adults will be enrolled in double blind manner.
  Interventions: Drug: TAK-925
- Part 1: Placebo (Cohort 1-2) (Placebo Comparator): TAK-925 Placebo, Intravenous single administration. Healthy adults will be enrolled in double blind manner.
  Interventions: Drug: Placebo
- Part 1: TAK-925 (Cohort 3; Dose Level 5) (Experimental): TAK-925, Intravenous single administration. Dose level will be determined by targeted plasma level of TAK-925 (Dose level 5). Healthy elderly participants will be enrolled in double blind manner.
  Interventions: Drug: TAK-925
- Part 1: Placebo (Cohort 3) (Placebo Comparator): TAK-925 Placebo, Intravenous single administration. Healthy elderly participants will be enrolled in double blind manner.
  Interventions: Drug: Placebo
- Part 1: TAK-925 (Cohort 4; Dose Level 5) (Experimental): TAK-925, Intravenous single administration. Dose level will be determined by targeted plasma level of TAK-925 (Dose level 5). Healthy adults will be enrolled in non-blinded manner.
  Interventions: Drug: TAK-925
- Part 2: TAK-925 TBD (Cohort 5) (Experimental): TAK-925, Intravenous single administration. Dose in Cohort 5 will be based on safety and tolerability in the Part 1. Patients with Narcolepsy will be enrolled in double blind manner (sponsor open).
  Interventions: Drug: TAK-925
- Part 2: TAK-925 TBD (Cohort 6) (Experimental): TAK-925, Intravenous single administration. Dose in Cohort 6 TBD based on safety, tolerability, PK data, and results of the Maintenance Wakefulness Test (MWT) from previous Cohorts. Patients with Narcolepsy will be enrolled in double blind manner (sponsor open).
  Interventions: Drug: TAK-925
- Part 2: TAK-925 TBD (Cohort 7) (Experimental): TAK-925, Intravenous single administration. Dose in Cohort 7 TBD based on safety, tolerability, PK data, and results of the Maintenance of Wakefulness Test (MWT) from previous Cohorts. Patients with Narcolepsy will be enrolled in double blind manner (sponsor open).
  Interventions: Drug: TAK-925
- Part 2: Placebo (Cohort 5-7) (Placebo Comparator): TAK-925 Placebo, Intravenous single administration. Patients with Narcolepsy will be enrolled in double blind manner (sponsor open).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-925 — TAK-925 Intravenous Infusion
  Arms: Part 1: TAK-925 (Cohort 1; Dose Level 1); Part 1: TAK-925 (Cohort 1; Dose Level 3); Part 1: TAK-925 (Cohort 1; Dose Level 5); Part 1: TAK-925 (Cohort 2; Dose Level 2); Part 1: TAK-925 (Cohort 2; Dose Level 4); Part 1: TAK-925 (Cohort 2; Dose Level 6); Part 1: TAK-925 (Cohort 3; Dose Level 5); Part 1: TAK-925 (Cohort 4; Dose Level 5); Part 2: TAK-925 TBD (Cohort 5); Part 2: TAK-925 TBD (Cohort 6); Part 2: TAK-925 TBD (Cohort 7)
Drug: Placebo — TAK-925 Placebo Intravenous Infusion
  Arms: Part 1: Placebo (Cohort 1-2); Part 1: Placebo (Cohort 3); Part 2: Placebo (Cohort 5-7)

SUMMARY:
The purpose of this study is to investigate safety, tolerability, and pharmacokinetics of TAK-925 when a single dose of TAK-925 is administered to healthy adult participants, healthy elderly participants and patients with type 1 narcolepsy.

DETAILED DESCRIPTION:
Orexins are neuropeptides that play a role in the regulation of sleep and wakefulness. In type 1 narcolepsy, there is a loss of orexin producing neurons in the brain. The investigational drug, TAK-925, is an orexin 2 receptor agonist that is being tested in healthy adult participants, healthy elderly participants and patients with narcolepsy in order to evaluate the safety, tolerability, and pharmacokinetics (PK) of a single intravenous administration.

The study will enroll approximately 20 healthy participants and 16 healthy elderly participants in Part 1 of the study and approximately 20 patients with narcolepsy in Part 2.

In Part 1, the study consists of 4 cohorts of 8 or 4 participants each. Participants will be randomly assigned (by chance, like flipping a coin) to one of the following treatment groups to receive TAK-925 or placebo:

- Part 1, Cohort 1; TAK-925 (Dose Level 1, 3, 5), Cohort 2; TAK-925 (Dose Level 2, 4, 6), Cohort 3 and 4; TAK-925 (Dose Level 5)

For Cohort 1-4, healthy adult and elderly participants will be administered TAK-925 or placebo once in each cohort or dose level. The dose at the start (Cohort 1 dose level 1) is 7 mg of TAK-925 and following doses in Cohorts 1-4 will be determined based on available data from previous Cohorts/dose levels.

In Part 2 of the study, the study consists of 3 cohorts of 4 to 12 patients with narcolepsy. Patients will be randomly assigned to one of the treatment groups of Cohort 5-7 and will be administered TAK-925 or placebo once in each cohort. The dose of TAK-925 in Cohort 5-7 is TBD and will be decided based on available data from Part 1 and previous Cohorts.

- Part 2, Cohort 5-7

This multi-center trial will be conducted in Japan. Participants will make multiple visits to the clinic. Visits in Part 1 will include a screening period (Day -28 to -2), Check-in on Day -1, Treatment period (Day 1 and 2), and follow-up visit on Day 7. In Part 2 of the study, the visits include a screening period (Day -42 to -2), Check-in on Day -1, Cross-over period (Day 1 to 4), and follow-up visit on Day 7.

ELIGIBILITY:
Inclusion Criteria:

Healthy adult participants and Healthy elderly participants:

- Participant weighs at least 50 kilogram (kg) (Healthy adults participants) / 40 kg (Healthy elderly participants) and has a body mass index (BMI) from 18.5 to 30 kilogram per square meter (kg/m^2), inclusive at Screening.

Narcolepsy patients:

* Patient weighs at least 40 kg inclusive at Screening.
* A diagnosis of narcolepsy Type 1, as defined by the International Classification of Sleep Disorders, Third Edition (ICSD-3).
* HLA narcolepsy test positivity.
* At Day -1, Epworth sleepiness scale (ESS) score greater than or equal to (>=) 10
* Blood pressure less than (<) 140 systolic and < 90 diastolic. The patient may have a history of hypertension and be on antihypertensive medication treatment as long as the BP meets these criteria.

Exclusion Criteria:

All Participants:

* Participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 2 years prior to the Screening visit.
* Past or current epilepsy, convulsion, tremor or the disorders of related symptoms.
* Has a lifetime history of major psychiatric disorder, such as major depressive disorder, bipolar disorder, or schizophrenia.

HV (only Cohort 4):

- Participant has had CSF collection performed within 14 days prior to check-in (Day -1).

Narcolepsy patients

* Medical disorder associated with excessive sleepiness other than narcolepsy (including sleep apnea syndrome).
* Excessive caffeine (greater than [>] 400 milligram per day [mg/day]) use one week prior to study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-11-04 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- Japan (3):
  - Sumida Hospital, Sumida-ku, Tokyo
  - Hakata Clinic, Fukuoka
  - PS Clinic, Fukuoka

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in Japan from 04 November 2017 to 04 September 2018.
Pre-assignment Details: Healthy adult and elderly participants were enrolled to receive TAK-925 or placebo in Cohorts 1 and 2 under alternating panel design and in Cohorts S1, S2, 3, and 4 under parallel design of Part 1, and participants with type 1 narcolepsy were enrolled to receive TAK-925 or placebo in a 2-period cross-over design in Cohorts 5, 6, and 7 of Part 2.
Groups:
- Part 1 Cohort 1: TAK-925 7 mg + TAK-925 28 mg + TAK-925 112 mg: TAK-925 7 milligram (mg), infusion, intravenously, once on Day 1 of Period 1, followed by TAK-925 28 mg infusion, intravenously, once on Day 1 of Period 2, further followed by TAK-925 112 mg infusion, intravenously, once on Day 1 of Period 3 in healthy adults in Group A in double-blind, alternating panel.
- Part 1 Cohort 1: TAK-925 7 mg + TAK-925 28 mg + Placebo: TAK-925 7 mg, infusion, intravenously, once on Day 1 of Period 1, followed by TAK-925 28 mg infusion, intravenously, once on Day 1 of Period 2, further followed by TAK-925 placebo-matching infusion, intravenously, once on Day 1 of Period 3 in healthy adults in Group B in double-blind, alternating panel.
- Part 1 Cohort 1: TAK-925 7 mg + Placebo + TAK-925 112 mg: TAK-925 7 mg, infusion, intravenously, once on Day 1 of Period 1, followed by TAK-925 placebo-matching infusion, intravenously, once on Day 1 of Period 2, further followed by TAK-925 112 mg, infusion, intravenously, once on Day 1 of Period 3 in healthy adults in Group C in double-blind, alternating panel.
- Part 1 Cohort 1: Placebo + TAK-925 28 mg + TAK-925 112 mg: TAK-925 placebo-matching infusion, intravenously, once on Day 1 of Period 1, followed by TAK-925 28 mg, infusion, intravenously, once on Day 1 of Period 2, further followed by TAK-925 112 mg, infusion, intravenously, once on Day 1 of Period 3 in healthy adults in Group D in double-blind, alternating panel.
- Part 1 Cohort 2:TAK-925 14 mg +TAK-925 56 mg +TAK-925 134.4 mg: TAK-925 14 mg, infusion, intravenously, once on Day 1 of Period 1, followed by TAK-925 56 mg infusion, intravenously, once on Day 1 of Period 2, further followed by TAK-925 134.4 mg infusion, intravenously, once on Day 1 of Period 3 in healthy adults in Group E in double-blind, alternating panel.
- Part 1 Cohort 2: TAK-925 14 mg + TAK-925 56 mg + Placebo: TAK-925 14 mg, infusion, intravenously, once on Day 1 of Period 1, followed by TAK-925 56 mg infusion, intravenously, once on Day 1 of Period 2, further followed by TAK-925 placebo-matching infusion, intravenously, once on Day 1 of Period 3 in Group F in healthy adults in double-blind, alternating panel.
- Part 1 Cohort 2: TAK-925 14 mg + Placebo + TAK-925 134.4 mg: TAK-925 14 mg, infusion, intravenously, once on Day 1 of Period 1, followed by TAK-925 placebo-matching infusion, intravenously, once on Day 1 of Period 2, further followed by TAK-925 134.4 mg infusion, intravenously, once on Day 1 of Period 3 in healthy adults in Group G in double-blind, alternating panel.
- Part 1 Cohort 2: Placebo + TAK-925 56 mg + TAK-925 134.4 mg: TAK-925 placebo-matching infusion, intravenously, once on Day 1 of Period 1, followed by TAK-925 56 mg infusion, intravenously, once on Day 1 of Period 2, further followed by TAK-925 134.4 mg infusion, intravenously, once on Day 1 of Period 3 in healthy adults in Group H in double-blind, alternating panel.
- Part 1 Cohort S1-S2: Pooled Placebo: TAK-925 placebo-matching infusion, intravenously, once on Day 1 in healthy adults in double-blind, parallel group.
- Part 1 Cohort S1: TAK-925 180 mg: TAK-925 180 mg, infusion, intravenously, once on Day 1 in healthy adults in double-blind, parallel group.
- Part 1 Cohort S2: TAK-925 240 mg: TAK-925 240 mg, infusion, intravenously, once on Day 1 in healthy adults in double-blind, parallel group.
- Part 1 Cohort 3: Placebo: TAK-925 placebo-matching infusion, intravenously, once on Day 1 in healthy elderly participants in double-blind, parallel group.
- Part 1 Cohort 3: TAK-925 112 mg: TAK-925 112 mg, infusion, intravenously, once on Day 1 in healthy elderly participants in double-blind, parallel group.
- Part 1 Cohort 4: TAK-925 112 mg: TAK-925 112 mg, infusion, intravenously, once on Day 1 in healthy adults in unblinded manner.
- Part 2 Cohort 5: TAK-925 44.8 mg + Placebo: TAK-925 44.8 mg, infusion, intravenously, once on Day 1 of Period 1, followed by TAK-925 placebo-matching infusion, intravenously, once on Day 1 of Period 2 (Day 3) in participants with type 1 narcolepsy in Group I under 2-period crossover design. A washout period of 7 days was required before the dosing on Day 1 for prior medications.
- Part 2 Cohort 5: Placebo + TAK-925 44.8 mg: TAK-925 placebo-matching infusion, intravenously, once on Day 1 of Period 1, followed by TAK-925 44.8 mg, infusion, intravenously, once on Day 1 of Period 2 (Day 3) in participants with type 1 narcolepsy in Group J under 2-period crossover design. A washout period of 7 days was required before the dosing on Day 1 for prior medications.
- Part 2 Cohort 6: TAK-925 11.2 mg + Placebo: TAK-925 11.2 mg, infusion, intravenously, once on Day 1 of Period 1, followed by TAK-925 placebo-matching infusion, intravenously, once on Day 1 of Period 2 (Day 3) in participants with type 1 narcolepsy in Group K under 2-period crossover design. A washout period of 7 days was required before the dosing on Day 1 for prior medications.
- Part 2 Cohort 6: Placebo + TAK-925 11.2 mg: TAK-925 placebo-matching infusion, intravenously, once on Day 1 of Period 1, followed by TAK-925 11.2 mg, infusion, intravenously, once on Day 1 Period 2 (Day 3) in participants with type 1 narcolepsy in Group L under 2-period crossover design. A washout period of 7 days was required before the dosing on Day 1 for prior medications.
- Part 2 Cohort 7: TAK-925 5 mg + Placebo: TAK-925 5 mg, infusion, intravenously, once on Day 1 of Period 1, followed by TAK-925 placebo-matching infusion, intravenously, once on Day 1 of Period 2 (Day 3) in participants with type 1 narcolepsy in Group M under 2-period crossover design. A washout period of 7 days was required before the dosing on Day 1 for prior medications.
- Part 2 Cohort 7: Placebo + TAK-925 5 mg: TAK-925 placebo-matching infusion, intravenously, once on Day 1 of Period 1, followed by TAK-925 5 mg, infusion, intravenously, once on Day 1 of Period 2 (Day 3) in participants with type 1 narcolepsy in Group N under 2-period crossover design. A washout period of 7 days was required before the dosing on Day 1 for prior medications
Period: Parts 1 and 2 - Period 1 (1 Day)
Arm/Group | Part 1 Cohort 1: TAK-925 7 mg + TAK-925 28 mg + TAK-925 112 mg | Part 1 Cohort 1: TAK-925 7 mg + TAK-925 28 mg + Placebo | Part 1 Cohort 1: TAK-925 7 mg + Placebo + TAK-925 112 mg | Part 1 Cohort 1: Placebo + TAK-925 28 mg + TAK-925 112 mg | Part 1 Cohort 2:TAK-925 14 mg +TAK-925 56 mg +TAK-925 134.4 mg | Part 1 Cohort 2: TAK-925 14 mg + TAK-925 56 mg + Placebo | Part 1 Cohort 2: TAK-925 14 mg + Placebo + TAK-925 134.4 mg | Part 1 Cohort 2: Placebo + TAK-925 56 mg + TAK-925 134.4 mg | Part 1 Cohort S1-S2: Pooled Placebo | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: Placebo | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg | Part 2 Cohort 5: TAK-925 44.8 mg + Placebo | Part 2 Cohort 5: Placebo + TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg + Placebo | Part 2 Cohort 6: Placebo + TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg + Placebo | Part 2 Cohort 7: Placebo + TAK-925 5 mg
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 4 | 6 | 6 | 2 | 6 | 4 | 2 (A washout period of 7 days was required before the dosing on Day 1 for prior medications.) | 2 (A washout period of 7 days was required before the dosing on Day 1 for prior medications.) | 2 (A washout period of 7 days was required before the dosing on Day 1 for prior medications.) | 2 (A washout period of 7 days was required before the dosing on Day 1 for prior medications.) | 3 (A washout period of 7 days was required before the dosing on Day 1 for prior medications.) | 3 (A washout period of 7 days was required before the dosing on Day 1 for prior medications.)
Completed | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 4 | 6 | 6 | 2 | 6 | 4 | 1 | 2 | 2 | 2 | 3 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Parts 1 and 2- Period 2 (1 Day)
Arm/Group | Part 1 Cohort 1: TAK-925 7 mg + TAK-925 28 mg + TAK-925 112 mg | Part 1 Cohort 1: TAK-925 7 mg + TAK-925 28 mg + Placebo | Part 1 Cohort 1: TAK-925 7 mg + Placebo + TAK-925 112 mg | Part 1 Cohort 1: Placebo + TAK-925 28 mg + TAK-925 112 mg | Part 1 Cohort 2:TAK-925 14 mg +TAK-925 56 mg +TAK-925 134.4 mg | Part 1 Cohort 2: TAK-925 14 mg + TAK-925 56 mg + Placebo | Part 1 Cohort 2: TAK-925 14 mg + Placebo + TAK-925 134.4 mg | Part 1 Cohort 2: Placebo + TAK-925 56 mg + TAK-925 134.4 mg | Part 1 Cohort S1-S2: Pooled Placebo | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: Placebo | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg | Part 2 Cohort 5: TAK-925 44.8 mg + Placebo | Part 2 Cohort 5: Placebo + TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg + Placebo | Part 2 Cohort 6: Placebo + TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg + Placebo | Part 2 Cohort 7: Placebo + TAK-925 5 mg
Started | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 0 (Part 1 Cohorts S1-2, 3, and 4 participants did not continue in subsequent periods after Period 1.) | 0 (Part 1 Cohorts S1-2, 3, and 4 participants did not continue in subsequent periods after Period 1.) | 0 (Part 1 Cohorts S1-2, 3, and 4 participants did not continue in subsequent periods after Period 1.) | 0 (Part 1 Cohorts S1-2, 3, and 4 participants did not continue in subsequent periods after Period 1.) | 0 (Part 1 Cohorts S1-2, 3, and 4 participants did not continue in subsequent periods after Period 1.) | 0 (Part 1 Cohorts S1-2, 3, and 4 participants did not continue in subsequent periods after Period 1.) | 1 | 2 | 2 | 2 | 3 | 3
Completed | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1- Period 3 (1 Day)
Arm/Group | Part 1 Cohort 1: TAK-925 7 mg + TAK-925 28 mg + TAK-925 112 mg | Part 1 Cohort 1: TAK-925 7 mg + TAK-925 28 mg + Placebo | Part 1 Cohort 1: TAK-925 7 mg + Placebo + TAK-925 112 mg | Part 1 Cohort 1: Placebo + TAK-925 28 mg + TAK-925 112 mg | Part 1 Cohort 2:TAK-925 14 mg +TAK-925 56 mg +TAK-925 134.4 mg | Part 1 Cohort 2: TAK-925 14 mg + TAK-925 56 mg + Placebo | Part 1 Cohort 2: TAK-925 14 mg + Placebo + TAK-925 134.4 mg | Part 1 Cohort 2: Placebo + TAK-925 56 mg + TAK-925 134.4 mg | Part 1 Cohort S1-S2: Pooled Placebo | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: Placebo | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg | Part 2 Cohort 5: TAK-925 44.8 mg + Placebo | Part 2 Cohort 5: Placebo + TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg + Placebo | Part 2 Cohort 6: Placebo + TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg + Placebo | Part 2 Cohort 7: Placebo + TAK-925 5 mg
Started | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 0 (Part 1 Cohorts S1-2, 3, and 4 participants did not continue in subsequent periods after Period 1.) | 0 (Part 1 Cohorts S1-2, 3, and 4 participants did not continue in subsequent periods after Period 1.) | 0 (Part 1 Cohorts S1-2, 3, and 4 participants did not continue in subsequent periods after Period 1.) | 0 (Part 1 Cohorts S1-2, 3, and 4 participants did not continue in subsequent periods after Period 1.) | 0 (Part 1 Cohorts S1-2, 3, and 4 participants did not continue in subsequent periods after Period 1.) | 0 (Part 1 Cohorts S1-2, 3, and 4 participants did not continue in subsequent periods after Period 1.) | 0 (Part 2 participants did not continue in subsequent periods after Period 2.) | 0 (Part 2 participants did not continue in subsequent periods after Period 2.) | 0 (Part 2 participants did not continue in subsequent periods after Period 2.) | 0 (Part 2 participants did not continue in subsequent periods after Period 2.) | 0 (Part 2 participants did not continue in subsequent periods after Period 2.) | 0 (Part 2 participants did not continue in subsequent periods after Period 2.)
Completed | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Groups:
- Part 1 Cohort 1: TAK-925 7 mg + TAK-925 28 mg + TAK-925 112 mg: TAK-925 7 mg, infusion, intravenously, once on Day 1 of Period 1, followed by TAK-925 28 mg infusion, intravenously, once on Day 1 of Period 2, further followed by TAK-925 112 mg infusion, intravenously, once on Day 1 of Period 3 in healthy adults in Group A in double-blind, alternating panel.
- Part 1: Cohort S1 TAK-925 180 mg: TAK-925 180 mg, infusion, intravenously, once, over 9 hours on Day 1 in healthy adults in double-blind, parallel group.
- Part 1: Cohort S2 TAK-925 240 mg: TAK-925 240 mg, infusion, intravenously, once, over 9 hours on Day 1 in healthy adults in double-blind, parallel group.
- Part 1: Cohort 3 Placebo: TAK-925 placebo-matching infusion, intravenously, once, over 9 hours on Day 1 in healthy elderly participants in double-blind, parallel group.
- Part 1: Cohort 3 TAK-925 112 mg: TAK-925 112 mg, infusion, intravenously, once, over 9 hours on Day 1 in healthy elderly participants in double-blind, parallel group.
- Part 1: Cohort 4 TAK-925 112 mg: TAK-925 112 mg, infusion, intravenously, once, over 9 hours on Day 1 in healthy adults in unblinded manner.
- Part 2 Cohort 5, Part J: TAK-925 Placebo + 44.8 mg: TAK-925 placebo-matching infusion, intravenously, once on Day 1 of Period 1, followed by TAK-925 44.8 mg, infusion, intravenously, once on Day 1 of Period 2 (Day 3) in participants with type 1 narcolepsy in Group J under 2-period crossover design. A washout period of 7 days was required before the dosing on Day 1 for prior medications.
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort 1: TAK-925 7 mg + TAK-925 28 mg + TAK-925 112 mg | Part 1 Cohort 1: TAK-925 7 mg + TAK-925 28 mg + Placebo | Part 1 Cohort 1: TAK-925 7 mg + Placebo + TAK-925 112 mg | Part 1 Cohort 1: Placebo + TAK-925 28 mg + TAK-925 112 mg | Part 1 Cohort 2:TAK-925 14 mg +TAK-925 56 mg +TAK-925 134.4 mg | Part 1 Cohort 2: TAK-925 14 mg + TAK-925 56 mg + Placebo | Part 1 Cohort 2: TAK-925 14 mg + Placebo + TAK-925 134.4 mg | Part 1 Cohort 2: Placebo + TAK-925 56 mg + TAK-925 134.4 mg | Part 1 Cohort S1-S2: Pooled Placebo | Part 1: Cohort S1 TAK-925 180 mg | Part 1: Cohort S2 TAK-925 240 mg | Part 1: Cohort 3 Placebo | Part 1: Cohort 3 TAK-925 112 mg | Part 1: Cohort 4 TAK-925 112 mg | Part 2 Cohort 5: TAK-925 44.8 mg + Placebo | Part 2 Cohort 5, Part J: TAK-925 Placebo + 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg + Placebo | Part 2 Cohort 6: Placebo + TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg + Placebo | Part 2 Cohort 7: Placebo + TAK-925 5 mg | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 4 | 6 | 6 | 2 | 6 | 4 | 2 | 2 | 2 | 2 | 3 | 3 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (5.66) | 25.5 (4.95) | 22.0 (2.83) | 30.0 (4.24) | 24.5 (3.54) | 28.0 (9.90) | 28.5 (9.19) | 34.5 (4.95) | 24.8 (4.57) | 24.5 (5.75) | 27.5 (6.72) | 72.5 (3.54) | 67.7 (2.94) | 21.3 (0.50) | 21.5 (4.95) | 33.0 (15.56) | 25.5 (7.78) | 38.5 (0.71) | 42.3 (20.11) | 33.7 (4.51) | 33.7 (16.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 0 | 0 | 2 | 3 | 1 | 12
  Male | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 4 | 6 | 6 | 1 | 3 | 4 | 0 | 2 | 2 | 0 | 0 | 2 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 4 | 6 | 6 | 2 | 6 | 4 | 2 | 2 | 2 | 2 | 3 | 3 | 58
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m˄2)] | 22.25 (2.475) | 22.35 (0.919) | 20.85 (2.899) | 22.10 (0.141) | 21.55 (2.616) | 20.90 (0.424) | 23.40 (2.687) | 22.15 (1.626) | 22.65 (1.912) | 20.48 (0.768) | 21.05 (1.325) | 23.00 (2.263) | 23.22 (3.451) | 22.03 (2.791) | 32.30 (10.041) | 24.60 (2.546) | 23.60 (0.707) | 26.45 (8.697) | 26.10 (7.146) | 29.57 (5.689) | 23.19 (4.072)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 176.0 (1.41) | 167.0 (2.83) | 174.5 (2.12) | 177.0 (8.49) | 170.0 (4.24) | 173.0 (1.41) | 170.0 (9.90) | 171.5 (6.36) | 173.5 (5.80) | 173.0 (3.16) | 168.8 (5.00) | 149.0 (0.00) | 159.5 (4.64) | 171.0 (5.89) | 155.5 (0.71) | 174.5 (6.36) | 171.0 (1.41) | 159.5 (2.12) | 160.7 (4.73) | 168.3 (11.55) | 168.1 (8.11)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 68.15 (7.707) | 62.65 (0.636) | 62.90 (10.607) | 69.60 (6.930) | 60.95 (5.445) | 62.45 (1.909) | 68.80 (14.849) | 63.85 (8.839) | 68.73 (1.941) | 61.12 (2.860) | 59.55 (6.142) | 51.30 (4.101) | 58.77 (10.388) | 63.88 (7.029) | 78.45 (24.112) | 74.95 (0.071) | 69.05 (1.202) | 67.70 (23.900) | 67.57 (22.212) | 83.43 (15.970) | 65.20 (10.994)
Smoking Classification [Count of Participants; unit: Participants]
  Non-smoker | 2 | 2 | 2 | 2 | 1 | 1 | 2 | 1 | 2 | 5 | 5 | 2 | 6 | 3 | 2 | 1 | 1 | 1 | 2 | 1 | 44
  Current smoker | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Former smoker | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 11
Alcohol Classification [Count of Participants; unit: Participants]
  Daily | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  A Few Times Per Week | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 10
  A Few Times Per Month | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 4 | 3 | 4 | 0 | 2 | 3 | 1 | 1 | 1 | 0 | 2 | 0 | 25
  Non-alcoholic | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 3 | 2 | 1 | 3 | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 22
Caffeine Classification [Count of Participants; unit: Participants]
  Had caffeine consumption | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 3 | 3 | 1 | 5 | 3 | 2 | 2 | 2 | 2 | 1 | 3 | 35
  Had no caffeine consumption | 0 | 2 | 2 | 0 | 2 | 1 | 1 | 1 | 3 | 3 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Time Frame: Baseline up to Day 7
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 Cohort 1-2: Pooled Placebo: TAK-925 placebo-matching infusion, intravenously, once on Day 1 in healthy adults in Group A to H in double-blind, alternating panel.
- Part 1 Cohort 1: TAK-925 7 mg: TAK-925 7 mg, infusion, intravenously, once on Day 1 in healthy adults in Group A to D in double-blind, alternating panel.
- Part 1 Cohort 2: TAK-925 14 mg: TAK-925 14 mg, infusion, intravenously, once on Day 1 in healthy adults in Group E to H in double-blind, alternating panel.
- Part 1 Cohort 1: TAK-925 28 mg: TAK-925 28 mg, infusion, intravenously, once on Day 1 in healthy adults in Group A to D in double-blind, alternating panel.
- Par 1 Cohort 2: TAK-925 56 mg: TAK-925 56 mg, infusion, intravenously, once on Day 1 in healthy adults in Group E to H in double-blind, alternating panel.
- Part 1 Cohort 1: TAK-925 112 mg: TAK-925 112 mg, infusion, intravenously, once on Day 1 in healthy adults in Group A to D in double-blind, alternating panel.
- Part 1 Cohort 2: TAK-925 134.4 mg: TAK-925 134.4 mg, infusion, intravenously, once on Day 1 in healthy adults in Group E to H in double-blind, alternating panel.
- Part 2 Cohort 5-7: Pooled Placebo: TAK-925 placebo-matching infusion, intravenously, once on Day 1 or Day 3 in participants with type 1 narcolepsy in Cohort 5 to 7 under 2-period crossover design.
- Part 2 Cohort 5: TAK-925 44.8 mg: TAK-925 44.8 mg, infusion, intravenously, once on Day 1 or Day 3 in participants with type 1 narcolepsy under 2-period crossover design.
- Part 2 Cohort 6: TAK-925 11.2 mg: TAK-925 11.2 mg, infusion, intravenously, once on Day 1 or Day 3 in participants with type 1 narcolepsy under 2-period crossover design.
- Part 2 Cohort 7: TAK-925 5 mg: TAK-925 5 mg, infusion, intravenously, once on Day 1 or Day 3 in participants with type 1 narcolepsy under 2-period crossover design.
Arm/Group | Part 1 Cohort 1-2: Pooled Placebo | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1-S2: Pooled Placebo | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: Placebo | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg | Part 2 Cohort 5-7: Pooled Placebo | Part 2 Cohort 5: TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg
Number analyzed (Participants) | 11 | 6 | 6 | 5 | 6 | 6 | 6 | 4 | 6 | 6 | 2 | 6 | 4 | 13 | 4 | 4 | 6
Participants | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 3 | 5 | 0 | 3 | 1 | 0 | 4 | 1 | 0

2. Primary Outcome: Number of Participants Who Experience at Least One TEAE Related to Vital Signs
Time Frame: Baseline up to Day 7
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1-2: Pooled Placebo | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1-S2: Pooled Placebo | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: Placebo | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg | Part 2 Cohort 5-7: Pooled Placebo | Part 2 Cohort 5: TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg
Number analyzed (Participants) | 11 | 6 | 6 | 5 | 6 | 6 | 6 | 4 | 6 | 6 | 2 | 6 | 4 | 13 | 4 | 4 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 4 | 0 | 3 | 0 | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants Who Experience at Least One TEAE Related to Body Weight
Time Frame: Baseline up to Day 7
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1-2: Pooled Placebo | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1-S2: Pooled Placebo | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: Placebo | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg | Part 2 Cohort 5-7: Pooled Placebo | Part 2 Cohort 5: TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg
Number analyzed (Participants) | 11 | 6 | 6 | 5 | 6 | 6 | 6 | 4 | 6 | 6 | 2 | 6 | 4 | 13 | 4 | 4 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Who Experience at Least One TEAE Related to 12-lead Electrocardiogram (ECG)
Time Frame: Baseline up to Day 7
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1-2: Pooled Placebo | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1-S2: Pooled Placebo | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: Placebo | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg | Part 2 Cohort 5-7: Pooled Placebo | Part 2 Cohort 5: TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg
Number analyzed (Participants) | 11 | 6 | 6 | 5 | 6 | 6 | 6 | 4 | 6 | 6 | 2 | 6 | 4 | 13 | 4 | 4 | 6
Participants | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Who Experience at Least One TEAE Related to Clinical Laboratory Tests
Time Frame: Baseline up to Day 7
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1-2: Pooled Placebo | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1-S2: Pooled Placebo | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: Placebo | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg | Part 2 Cohort 5-7: Pooled Placebo | Part 2 Cohort 5: TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg
Number analyzed (Participants) | 11 | 6 | 6 | 5 | 6 | 6 | 6 | 4 | 6 | 6 | 2 | 6 | 4 | 13 | 4 | 4 | 6
Participants | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part 1, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-925 and Its Metabolites M1 and M2
Time Frame: Day 1 pre-infusion and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 9 hours after the start of infusion and at 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 10 and 15 hours post-infusion
Population: The PK analysis set was defined as all participants who received at least one dose of study drug and whose plasma or cerebrospinal fluid (CSF) concentration was measured at least once or whose cumulative urinary excretion was calculated. Here "number analyzed" were participants who were evaluable for the outcome measure at given time points.
Measure: Geometric Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
hour*nanogram per milliliter (h*ng/mL)
  TAK-925: number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  TAK-925 | 138.0 (22.546) | 323.1 (45.793) | 513.3 (81.392) | 1055 (178.49) | 2069 (298.89) | 2655 (495.32) | 2994 (164.73) | 4542 (698.25) | 2546 (274.48) | 2011 (195.00)
  Metabolite M1: number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  Metabolite M1 | 74.10 (31.837) | 170.7 (50.607) | 293.1 (120.91) | 613.8 (218.79) | 1272 (409.93) | 1724 (596.04) | 1762 (204.30) | 3094 (740.81) | 1037 (343.80) | 996.3 (321.79)
  Metabolite M2: number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  Metabolite M2 | 0.3676 (0.89268) | 1.940 (2.5750) | 5.893 (2.8201) | 9.225 (6.3231) | 22.79 (19.464) | 31.23 (25.058) | 28.69 (4.9460) | 56.79 (21.993) | 15.96 (9.4609) | 16.81 (8.7980)

7. Primary Outcome: Part 2, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-925 and Its Metabolites M1 and M2
Time Frame: Days 1-4 pre-infusion and at 1, 2, 4, 6 and 9 hours after the start of infusion and at 0.17, 0.5, 1, 2 and 15 hours post-infusion
Population: The PK analysis set was defined as all participants who received at least one dose of study drug and whose plasma or CSF concentration was measured at least once or whose cumulative urinary excretion was calculated. Here "number analyzed" were participants who were evaluable for the outcome measure at given time points.
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 2 Cohort 5: TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg
Number analyzed (Participants) | 4 | 4 | 6
h*ng/mL
  TAK-925: number analyzed (Participants) | 4 | 4 | 4
  TAK-925 | 910.8 (275.10) | 198.7 (13.540) | 86.15 (14.777)
  Metabolite M1: number analyzed (Participants) | 4 | 4 | 5
  Metabolite M1 | 623.6 (516.16) | 100.7 (55.904) | 52.25 (17.041)
  Metabolite M2: number analyzed (Participants) | 4 | 2 | 0
  Metabolite M2 | 10.90 (22.384) | 3.435 (2.0430) |

8. Primary Outcome: Part 1, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-925 and Its Metabolites M1 and M2
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
h*ng/mL
  TAK-925: number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  TAK-925 | 141.8 (22.744) | 328.1 (51.138) | 523.5 (88.288) | 1065 (187.70) | 2092 (319.85) | 2682 (519.45) | 3013 (160.21) | 4585 (689.28) | 2590 (283.03) | 2028 (196.21)
  Metabolite M1: number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  Metabolite M1 | 75.77 (32.409) | 173.5 (53.475) | 296.1 (122.50) | 618.9 (221.98) | 1284 (409.94) | 1737 (606.78) | 1764 (202.65) | 3112 (745.48) | 1052 (350.05) | 1001 (323.04)
  Metabolite M2: number analyzed (Participants) | 1 | 4 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  Metabolite M2 | 2.900 | 5.302 (1.6898) | 6.416 (1.0512) | 9.796 (6.6369) | 23.79 (19.535) | 32.29 (25.766) | 29.43 (5.0744) | 57.72 (21.853) | 16.88 (9.9205) | 17.22 (8.8861)

9. Primary Outcome: Part 2, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-925 and Its Metabolites M1 and M2
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 2 Cohort 5: TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg
Number analyzed (Participants) | 4 | 4 | 6
h*ng/mL
  TAK-925: number analyzed (Participants) | 4 | 4 | 4
  TAK-925 | 925.3 (296.03) | 200.7 (13.216) | 88.45 (13.682)
  Metabolite M1: number analyzed (Participants) | 4 | 4 | 5
  Metabolite M1 | 634.0 (549.20) | 102.4 (55.929) | 54.77 (17.148)
  Metabolite M2: number analyzed (Participants) | 2 | 2 | 0
  Metabolite M2 | 27.99 (28.284) | 3.816 (0.60811) |

10. Primary Outcome: Part 1, Cmax: Maximum Observed Plasma Concentration for TAK-925 and Its Metabolites M1 and M2
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
nanogram per milliliter (ng/mL)
  TAK-925: number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  TAK-925 | 16.70 (2.8896) | 36.83 (4.3976) | 57.56 (8.2309) | 122.6 (13.014) | 235.2 (40.712) | 304.9 (50.702) | 344.5 (23.549) | 506.3 (87.027) | 278.4 (33.127) | 237.8 (25.695)
  Metabolite M1: number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  Metabolite M1 | 8.458 (3.5972) | 19.50 (4.9426) | 31.82 (11.983) | 67.69 (20.931) | 134.1 (45.828) | 189.2 (60.185) | 197.8 (26.011) | 333.2 (70.509) | 106.7 (30.612) | 114.4 (38.575)
  Metabolite M2: number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  Metabolite M2 | 0.2379 (0.11806) | 0.4290 (0.24813) | 0.7051 (0.33672) | 1.076 (0.63619) | 2.564 (2.0370) | 3.422 (2.4880) | 3.279 (0.53902) | 6.611 (2.2350) | 1.751 (0.90125) | 2.022 (0.99882)

11. Primary Outcome: Part 2, Cmax: Maximum Observed Plasma Concentration for TAK-925 and Its Metabolites M1 and M2
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2 Cohort 5: TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg
Number analyzed (Participants) | 4 | 4 | 6
ng/mL
  TAK-925: number analyzed (Participants) | 4 | 4 | 5
  TAK-925 | 96.48 (21.981) | 21.86 (2.5303) | 10.10 (1.9527)
  Metabolite M1: number analyzed (Participants) | 4 | 4 | 5
  Metabolite M1 | 64.28 (39.990) | 11.23 (5.0467) | 5.990 (1.8931)
  Metabolite M2: number analyzed (Participants) | 4 | 2 | 0
  Metabolite M2 | 1.305 (1.9483) | 0.4884 (0.28306) |

12. Primary Outcome: Part 1, Ceoi: Concentration at the End of Infusion for TAK-925 and Its Metabolites M1 and M2
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
ng/mL
  TAK-925: number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  TAK-925 | 13.37 (2.0174) | 29.81 (4.2579) | 52.08 (7.2344) | 114.6 (13.303) | 213.8 (31.714) | 290.3 (32.096) | 324.0 (30.182) | 493.2 (70.335) | 272.2 (36.985) | 183.5 (15.875)
  Metabolite M1: number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  Metabolite M1 | 7.532 (3.4019) | 17.79 (4.9179) | 28.06 (11.208) | 58.79 (23.607) | 121.3 (37.632) | 167.5 (58.242) | 174.0 (20.376) | 295.5 (75.002) | 98.82 (31.862) | 105.0 (38.567)
  Metabolite M2: number analyzed (Participants) | 3 | 6 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  Metabolite M2 | 0.2289 (0.12885) | 0.3978 (0.23853) | 0.5928 (0.27538) | 0.9225 (0.54081) | 2.217 (1.6608) | 3.079 (2.3329) | 2.850 (0.52592) | 4.868 (2.3897) | 1.528 (0.87452) | 1.624 (0.96722)

13. Primary Outcome: Part 2, Ceoi: Concentration at the End of Infusion for TAK-925 and Its Metabolites M1 and M2
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2 Cohort 5: TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg
Number analyzed (Participants) | 4 | 4 | 6
ng/mL
  TAK-925: number analyzed (Participants) | 4 | 4 | 5
  TAK-925 | 94.04 (23.643) | 21.17 (1.7896) | 9.649 (1.1339)
  Metabolite M1: number analyzed (Participants) | 4 | 4 | 5
  Metabolite M1 | 58.61 (42.471) | 9.916 (5.6434) | 5.412 (1.7517)
  Metabolite M2: number analyzed (Participants) | 4 | 2 | 0
  Metabolite M2 | 1.075 (1.8500) | 0.4037 (0.23357) |

14. Primary Outcome: Part 1, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-925 and Its Metabolites M1 and M2
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
hours
  TAK-925: number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  TAK-925 | 3.000 [2.00 to 4.00] | 4.000 [3.00 to 4.00] | 3.000 [2.00 to 4.00] | 4.000 [3.00 to 9.00] | 4.000 [1.50 to 9.00] | 6.500 [3.00 to 9.00] | 6.500 [3.00 to 9.00] | 4.000 [3.00 to 9.00] | 6.500 [1.50 to 9.00] | 5.000 [3.00 to 6.00]
  Metabolite M1: number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  Metabolite M1 | 6.000 [6.00 to 9.00] | 6.000 [6.00 to 9.00] | 6.000 [6.00 to 8.00] | 6.000 [6.00 to 9.00] | 6.000 [6.00 to 9.00] | 6.000 [6.00 to 8.00] | 6.000 [6.00 to 6.00] | 6.000 [6.00 to 6.00] | 6.000 [6.00 to 6.000] | 8.000 [8.00 to 8.00]
  Metabolite M2: number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  Metabolite M2 | 7.500 [4.00 to 9.00] | 8.000 [6.00 to 9.00] | 4.000 [4.00 to 4.00] | 6.000 [4.00 to 9.00] | 4.000 [3.00 to 6.00] | 4.000 [4.00 to 8.00] | 5.000 [4.00 to 6.00] | 3.500 [3.00 to 6.00] | 3.000 [1.50 to 9.00] | 3.500 [1.50 to 8.00]

15. Primary Outcome: Part 2, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-925 and Its Metabolites M1 and M2
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2 Cohort 5: TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg
Number analyzed (Participants) | 4 | 4 | 6
hours
  TAK-925: number analyzed (Participants) | 4 | 4 | 5
  TAK-925 | 6.500 [4.00 to 9.00] | 9.000 [4.00 to 9.00] | 9.000 [4.00 to 9.00]
  Metabolite M1: number analyzed (Participants) | 4 | 4 | 5
  Metabolite M1 | 6.000 [6.00 to 9.00] | 6.000 [6.00 to 9.00] | 6.000 [6.00 to 6.00]
  Metabolite M2: number analyzed (Participants) | 4 | 2 | 0
  Metabolite M2 | 5.960 [4.00 to 9.00] | 5.990 [5.98 to 6.00] |

16. Primary Outcome: Part 1, t1/2z: Terminal Disposition Phase Half-life of TAK-925 and Its Metabolites M1 and M2
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
hours
  TAK-925: number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  TAK-925 | 4.120 (1.9190) | 4.498 (1.7725) | 5.142 (1.8060) | 3.860 (0.6478) | 3.788 (1.0424) | 3.943 (0.9492) | 3.363 (0.8523) | 4.033 (1.2843) | 4.345 (0.5901) | 4.490 (1.5939)
  Metabolite M1: number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  Metabolite M1 | 2.598 (1.3239) | 3.443 (0.9386) | 3.122 (0.4673) | 2.760 (0.8950) | 3.075 (0.5984) | 2.825 (0.5203) | 2.205 (0.2616) | 2.637 (0.5575) | 3.763 (0.7675) | 2.400 (0.6307)
  Metabolite M2: number analyzed (Participants) | 1 | 4 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  Metabolite M2 | 2.670 | 1.8975 (0.2583) | 1.545 (0.1237) | 1.692 (0.7082) | 2.158 (0.7646) | 2.847 (1.5995) | 1.702 (0.4891) | 2.818 (1.0856) | 2.727 (1.3977) | 1.205 (0.2873)

17. Primary Outcome: Part 2, t1/2z: Terminal Disposition Phase Half-life of TAK-925 and Its Metabolites M1 and M2
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 2 Cohort 5: TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg
Number analyzed (Participants) | 4 | 4 | 6
hours
  TAK-925: number analyzed (Participants) | 4 | 4 | 4
  TAK-925 | 4.130 (1.1981) | 3.923 (1.0265) | 3.465 (1.0998)
  Metabolite M1: number analyzed (Participants) | 4 | 4 | 5
  Metabolite M1 | 3.670 (0.9131) | 2.523 (1.0892) | 2.154 (0.4215)
  Metabolite M2: number analyzed (Participants) | 2 | 2 | 0
  Metabolite M2 | 4.120 (2.5032) | 0.915 (0.2192) |

18. Primary Outcome: Part 1, Vss: Volume of Distribution at Steady State After Intravenous Administration for TAK-925
Time Frame: as for outcome 6
Population: The PK analysis set was defined as all participants who received at least one dose of study drug and whose plasma or CSF concentration was measured at least once or whose cumulative urinary excretion was calculated. Here "overall participants analyzed" are participants who were available for this outcome measure assessment at given time period.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg
Number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
liter | 82.88 (29.543) | 77.07 (22.804) | 116.1 (35.215) | 91.40 (14.122) | 97.83 (22.194) | 88.47 (12.476) | 90.75 (24.140) | 97.48 (28.378) | 99.48 (15.472) | 77.98 (28.931)

19. Primary Outcome: Part 2, Vss: Volume of Distribution at Steady State After Intravenous Administration for TAK-925
Time Frame: as for outcome 7
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Part 2 Cohort 5: TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg
Number analyzed (Participants) | 4 | 4 | 4
liter | 116.8 (7.8049) | 114.1 (14.964) | 111.7 (26.464)

20. Primary Outcome: Part 1, Vz: Volume of Distribution During the Terminal Phase After Intravenous Administration for TAK-925
Time Frame: as for outcome 6
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg
Number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
liter | 292.2 (124.03) | 271.7 (79.238) | 391.8 (117.09) | 290.7 (31.156) | 288.8 (55.185) | 284.7 (65.265) | 290.8 (77.783) | 313.0 (128.81) | 271.5 (39.145) | 357.3 (121.15)

21. Primary Outcome: Part 2, Vz: Volume of Distribution During the Terminal Phase After Intravenous Administration for TAK-925
Time Frame: as for outcome 7
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Part 2 Cohort 5: TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg
Number analyzed (Participants) | 4 | 4 | 4
liter | 281.3 (35.855) | 316.8 (84.263) | 282.3 (88.729)

22. Primary Outcome: Part 1, CL: Total Clearance After Intravenous Administration for TAK-925
Time Frame: as for outcome 6
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Arm/Group | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg
Number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
liter per hour (L/h) | 50.00 (9.0785) | 43.07 (6.4856) | 54.20 (9.9541) | 53.10 (8.2202) | 54.10 (9.0437) | 50.90 (9.8018) | 59.83 (3.3381) | 52.78 (7.4882) | 43.50 (4.9651) | 55.40 (5.2211)

23. Primary Outcome: Part 2, CL: Total Clearance After Intravenous Administration for TAK-925
Time Frame: as for outcome 7
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part 2 Cohort 5: TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg
Number analyzed (Participants) | 4 | 4 | 4
L/h | 50.18 (15.533) | 55.90 (3.7692) | 57.05 (9.5577)

24. Primary Outcome: Part 1, Ae(0-24): Amount of TAK-925 and Its Metabolites M1 and M2 Excreted in Urine From Time 0 to Time 24
Description: Urine assessments were done only in Part 1, as planned.
Time Frame: Day 1 pre-infusion and 0-9 hours after the start of infusion and at 0-3, 3-6, 6-15 and 15-24 hours post-infusion
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: microgram (mcg)
Arm/Group | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg
Number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
microgram (mcg)
  TAK-925 | 1.892 (0.93889) | 5.460 (3.4291) | 14.10 (2.4515) | 60.87 (23.008) | 210.5 (75.775) | 335.8 (117.81) | 578.5 (110.30) | 1223 (76.855) | 214.3 (137.61) | 184.8 (53.662)
  Metabolite M1 | 198.8 (49.600) | 426.7 (101.25) | 792.8 (253.36) | 1697 (495.32) | 1905 (1490.9) | 5228 (1785.9) | 5815 (1095.4) | 8163 (945.57) | 2343 (635.69) | 3193 (677.37)
  Metabolite M2 | 0.000 (0.0000) | 1.152 (1.5202) | 2.438 (2.2612) | 8.695 (5.3533) | 31.25 (26.282) | 40.08 (28.904) | 43.12 (8.4203) | 79.90 (23.679) | 14.37 (6.0079) | 21.01 (10.331)

25. Primary Outcome: Part 1, Fe(0-24): Fraction of Administered Dose of Drug Excreted in Urine From Time 0 to Time 24 for TAK-925 and Its Metabolites M1 and M2
Description: Urine assessments were done only in Part 1, as planned.
Time Frame: Day 1 pre-infusion and 0-9 hours after the start of infusion and at 0-3, 3-6, 6-15 and 15-24 hours post-infusion
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg
Number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
percentage of dose
  TAK-925 | 0.028 (0.0148) | 0.038 (0.0232) | 0.050 (0.0071) | 0.110 (0.0424) | 0.190 (0.0657) | 0.250 (0.0883) | 0.322 (0.0624) | 0.508 (0.0319) | 0.192 (0.1237) | 0.165 (0.0480)
  Metabolite M1 | 2.736 (0.6841) | 2.938 (0.6950) | 2.726 (0.8677) | 2.920 (0.8519) | 3.358 (1.2922) | 3.748 (1.2809) | 3.112 (0.5872) | 3.280 (0.3788) | 2.015 (0.5452) | 2.748 (0.5871)
  Metabolite M2 | 0.000 (0.0000) | 0.008 (0.0117) | 0.008 (0.0084) | 0.017 (0.0103) | 0.025 (0.0243) | 0.028 (0.0214) | 0.023 (0.0052) | 0.032 (0.0117) | 0.013 (0.0082) | 0.018 (0.0096)

26. Primary Outcome: Part 1, CLR: Renal Clearance of TAK-925 and Its Metabolites M1 and M2
Description: Urine assessments were done only in Part 1, as planned.
Time Frame: Day 1 pre-infusion and 0-9 hours after the start of infusion and at 0-3, 3-6 and 6-15 hours post-infusion
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
L/h
  TAK-925: number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  TAK-925 | 0.01390 (0.0071503) | 0.01656 (0.0097578) | 0.02746 (0.0053337) | 0.05672 (0.018842) | 0.1020 (0.037350) | 0.1275 (0.046864) | 0.1928 (0.035244) | 0.2705 (0.031501) | 0.08337 (0.053779) | 0.09053 (0.018093)
  Metabolite M1: number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  Metabolite M1 | 2.664 (0.83930) | 2.438 (0.30142) | 2.614 (0.54500) | 2.653 (0.24138) | 2.952 (0.65615) | 2.878 (0.35459) | 3.285 (0.49152) | 2.643 (0.37012) | 2.205 (0.35172) | 3.173 (0.50684)
  Metabolite M2: number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 4
  Metabolite M2 | 0.000 (0.0000) | 0.2182 (0.25950) | 0.4630 (0.31605) | 0.7897 (0.077544) | 1.014 (0.23516) | 1.041 (0.12104) | 1.468 (0.20508) | 1.353 (0.12894) | 0.7967 (0.15368) | 1.132 (0.24401)

27. Primary Outcome: Part 1, R(CSF/Plasma,ss): Cerebrospinal Fluid/Plasma Drug Concentration at Steady State for TAK-925 and Its Metabolites M1 and M2 in Cohort 4
Time Frame: Day 1 at 6 hours after start of infusion
Population: The PK analysis set was defined as all participants who received at least one dose of study drug and whose plasma or CSF concentration was measured at least once or whose cumulative urinary excretion was calculated.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1 Cohort 4: TAK-925 112 mg
Number analyzed (Participants) | 4
Ratio
  TAK-925 | 0.02848 (0.0056258)
  Metabolite M1 | 0.06190 (0.010358)
  Metabolite M2 | 0.02818 (0.032718)

28. Secondary Outcome: Part 2: Average Sleep Latency in Maintenance of Wakefulness Test (MWT)
Description: The MWT is a validated objective measure that evaluates a person's ability to remain awake under soporific conditions for a defined period of time. This tendency to fall asleep is measured via electroencephalography-derived sleep latency. Sleep onset is defined as the first epoch of greater than 15 seconds of cumulative sleep in a 30-second epoch. Trials were ended after 40 minutes if no sleep occurs, or after unequivocal sleep, defined as 3 consecutive epochs of stage 1 sleep, or 1 epoch of any other stage of sleep. If no sleep has been observed according to these rules, then the latency is defined as 40 minutes. MWT sleep latency ranges from 0 to 40 minutes, with higher scores indicating greater ability to stay awake.
Time Frame: Days 1 and 3 up to 8 hours following the start of infusion
Population: The pharmacodynamic analysis set was defined as all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part 2 Cohort 5-7: Pooled Placebo | Part 2 Cohort 5: TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg
Number analyzed (Participants) | 13 | 4 | 4 | 6
minutes | 2.88 (1.646) | 40.00 (0.000) | 37.59 (4.813) | 22.38 (10.125)
Statistical Analysis 1: Comparison: Part 2 Cohort 5-7: Pooled Placebo vs Part 2 Cohort 5: TAK-925 44.8 mg; Test type: Superiority; p < 0.0001, ANOVA — The p-value for each treatment group is for the comparison of that treatment group to the placebo treatment group
Statistical Analysis 2: Comparison: Part 2 Cohort 5-7: Pooled Placebo vs Part 2 Cohort 6: TAK-925 11.2 mg; Test type: Superiority; p < 0.0001, ANOVA — The p-value for each treatment group is for the comparison of that treatment group to the placebo treatment group
Statistical Analysis 3: Comparison: Part 2 Cohort 5-7: Pooled Placebo vs Part 2 Cohort 7: TAK-925 5 mg; Test type: Superiority; p = 0.0001, ANOVA — The p-value for each treatment group is for the comparison of that treatment group to the placebo treatment group

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 7 days (Day 7) after the last dose of study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1 Cohort 1-2: Pooled Placebo | Part 1 Cohort 1: TAK-925 7 mg | Part 1 Cohort 2: TAK-925 14 mg | Part 1 Cohort 1: TAK-925 28 mg | Par 1 Cohort 2: TAK-925 56 mg | Part 1 Cohort 1: TAK-925 112 mg | Part 1 Cohort 2: TAK-925 134.4 mg | Part 1 Cohort S1-S2: Pooled Placebo | Part 1 Cohort S1: TAK-925 180 mg | Part 1 Cohort S2: TAK-925 240 mg | Part 1 Cohort 3: Placebo | Part 1 Cohort 3: TAK-925 112 mg | Part 1 Cohort 4: TAK-925 112 mg | Part 2 Cohort 5-7: Pooled Placebo | Part 2 Cohort 5: TAK-925 44.8 mg | Part 2 Cohort 6: TAK-925 11.2 mg | Part 2 Cohort 7: TAK-925 5 mg
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/4 | 0/6 | 0/6 | 0/2 | 0/6 | 0/4 | 0/13 | 0/4 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/4 | 0/6 | 0/6 | 0/2 | 0/6 | 0/4 | 0/13 | 0/4 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 1/11 | 1/6 | 1/6 | 1/5 | 1/6 | 1/6 | 2/6 | 1/4 | 3/6 | 5/6 | 0/2 | 3/6 | 1/4 | 0/13 | 4/4 | 1/4 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohort 1-2: Pooled Placebo (N=11) | Part 1 Cohort 1: TAK-925 7 mg (N=6) | Part 1 Cohort 2: TAK-925 14 mg (N=6) | Part 1 Cohort 1: TAK-925 28 mg (N=5) | Par 1 Cohort 2: TAK-925 56 mg (N=6) | Part 1 Cohort 1: TAK-925 112 mg (N=6) | Part 1 Cohort 2: TAK-925 134.4 mg (N=6) | Part 1 Cohort S1-S2: Pooled Placebo (N=4) | Part 1 Cohort S1: TAK-925 180 mg (N=6) | Part 1 Cohort S2: TAK-925 240 mg (N=6) | Part 1 Cohort 3: Placebo (N=2) | Part 1 Cohort 3: TAK-925 112 mg (N=6) | Part 1 Cohort 4: TAK-925 112 mg (N=4) | Part 2 Cohort 5-7: Pooled Placebo (N=13) | Part 2 Cohort 5: TAK-925 44.8 mg (N=4) | Part 2 Cohort 6: TAK-925 11.2 mg (N=4) | Part 2 Cohort 7: TAK-925 5 mg (N=6)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling drunk (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 2 | 4 | 0 | 3 | 0 | 0 | 1 | 0 | 0
Electrocardiogram PR prolongation (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Narcolepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypnagogic hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Logorrhoea (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT03332784/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT03332784/SAP_001.pdf